CLINICAL TRIAL: NCT03855995
Title: A Prospective Study to Evaluate the Safety, Effectiveness and Impact of the RTS, S/AS01E Vaccine in Young Children in Sub-Saharan Africa
Brief Title: A Study Assessing the Safety, Efficacy, and Impact of GlaxoSmithKline Biologicals' RTS, S/AS01E Malaria Vaccine in Young Children Across Sub-Saharan Africa
Acronym: EPI-MAL-003
Status: Active, not recruiting | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115056
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Malaria; Malaria Vaccines
Keywords: Malaria; Plasmodium falciparum; Vaccine effectiveness; Sub-Saharan Africa; Active surveillance
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Cerebrospinal fluid

GROUPS / COHORTS (3):
- Active surveillance (DTP sub-Group): Children enrolled in the active surveillance (AS), <18 months of age who were identified at any administration of DTP/HepB/Hib (usually given at 6, 10 and 14 weeks of age) or at hospitalisation before administration of 3rd dose of DTP/HepB/Hib and vaccinated with at least one dose of DTP/HepB/Hib; including both RTS,S/AS01E vaccinated and unvaccinated children (from exposed or unexposed clusters), living in the HDSS area are eligible for enrolment in the DTP sub-group of active surveillance.
  Interventions: Procedure: Whole blood sample
- Active surveillance (Catch-up sub-Group): Children enrolled in the active surveillance (AS), <18 months of age who were identified at 1st RTS,S/AS01E dose administration and who either received all DTP/HepB/Hib doses before study start or received at least one dose of DTP/HepB/Hib and are older than the age corresponding to the 3rd DTP/HepB/Hib dose at study start; including only RTS,S/AS01E vaccinated children from exposed clusters who could not be recruited at the time of DTP/HepB/Hib administration because the study had not yet started, living in the HDSS area are eligible for enrolment in the Catch-up sub-group of active surveillance.
  Interventions: Procedure: Whole blood sample
- Enhanced Hospitalisation Surveillance Group: Children at least 6 weeks and <5 years of age, within the study areas in both exposed and unexposed clusters, not already enrolled in the active surveillance (because parents/ Legally Acceptable Representative (LARs) declined enrolment in active surveillance or because recruitment had been completed) or not eligible for active surveillance at the time of hospitalisation, living in the HDSS area are eligible for enrolment in the Enhanced Hospital Surveillance (EHS) group.
  Interventions: Procedure: Whole blood sample

INTERVENTIONS:
Procedure: Whole blood sample — Whole blood samples will be collected from all enrolled children hospitalised and suspected of having an AESI or meningitis.

SUMMARY:
The RTS, S/AS01E vaccine was developed to protect children in sub-Saharan Africa from malaria as part of routine immunization programs. This study aims to check the vaccine's safety after it has been introduced. Along with safety, researchers will also assess how well the vaccine works and its overall impact on children's health.

DETAILED DESCRIPTION:
This is a disease surveillance study with prospective cohort event monitoring including both temporal and concurrent comparisons of the occurrence of adverse and malaria events between vaccinated and unvaccinated subjects living in exposed or unexposed clusters located in sub-Saharan Africa (SSA) countries, and eligible for RTS,S/AS01E vaccination for those living in the exposed clusters. The design includes active surveillance and enhanced hospitalization surveillance in both exposed and unexposed clusters.

The study targeted enrolling at least 45,000 children in active surveillance, including 22,500 in the exposed clusters and 22,500 in the unexposed clusters for evaluation of the vaccine safety, effectiveness, and impact.

All data analyses will be computed in a descriptive manner. Data regarding the hospitalization will be uniformly collected whether the child is enrolled in active surveillance or in enhanced hospitalization surveillance.

ELIGIBILITY:
Inclusion Criteria

All study participants must satisfy ALL the following criteria at study entry:

* Study participants' parent(s)/ LAR(s) who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent provided from either the parent(s) or LAR of the study participant.
* Study participant living in the HDSS or equivalent surveillance system area.
* For enrolment in the active surveillance - DTP group: children must be aged less than (<) 18 months, identified at any administration of DTP/HepB/Hib (or at hospitalisation before 3rd dose of DTP/HepB/Hib in case of hospitalisation and vaccinated with at least one dose of DTP/HepB/Hib). (This group will include children from exposed and unexposed clusters.) OR For enrolment in the active surveillance - Catch-up group: children must be aged <18 months, received at least one dose of DTP/HepB/Hib vaccine, whose age corresponds to the age after the 3rd dose of DTP/HepB/Hib vaccine, (=who either received all DTP/HepB/Hib doses before study start or received at least one dose of DTP/HepB/Hib and are older than the age corresponding to the 3rd DTP/HepB/Hib dose at study start) and identified at 1st RTS,S/AS01E dose administration (This group will include children from exposed clusters only).

OR For enrolment in the enhanced hospitalisation surveillance: children must be aged at least 6 weeks and <5 years at the time of hospitalisation at any time during the study. (This group will include children from exposed and unexposed clusters.) Parents/LARs of children meeting all eligibility criteria for active surveillance, not having completed the visits for DTP/HepB/Hib, and first identified during hospitalisation, must first be proposed enrolment in active surveillance (if recruitment is not completed).

Children already enrolled in active surveillance will have hospitalization monitored as part of the procedures related to the active surveillance and can therefore not be enrolled in enhanced hospitalization surveillance.

Exclusion Criteria:

• Child in care = A child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government, or a government body, acting in accordance with powers conferred on them by law or regulation. The definition of a child in care can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a child in care does not include a child who is adopted or has an appointed legal guardian.

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The target population for the introduction of the RTS,S/AS01E vaccine are children living in the SSA.
Sampling Method: Probability Sample
Enrollment: 77969 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2025-08-11 (Estimated); Study Completion 2025-08-11 (Estimated)

PRIMARY OUTCOMES:
Incidence rates of adverse events of special interest (AESI) | During the entire study period (From Day 0 up to Month 62)
  AESI are predefined list of adverse events that have historically been associated with vaccines other than RTS,S/AS01E, or may hypothetically be associated with RTS,S/AS01E due to the fact that this vaccine has components which are new compared to current widely used vaccines.
  The incidence rate will be calculated by dividing the number of study participants reporting at least one event over the follow-up period by the total person-time. The person-time for an event of interest will be calculated as the time between the reference date (date of first RTS,S/AS01E vaccination for the vaccinated study participants and virtual vaccination corresponding to the week before first visit for the unvaccinated study participants) and the end of the at-risk period or the earliest of the followings: Date of first diagnosis of event of interest, Date of end of study period, Date when child reaches 5 years, Date of last contact or Date of death.
Incidence rates of aetiology-confirmed meningitis | During the entire study period (From Day 0 up to Month 62)
  Incidence rate of aetiology confirmed meningitis is analyzed with an at-risk period of 12 months. At the site level, a suspected meningitis case based on clinical symptoms and/or signs is defined as:
  * A child with sudden onset of fever (> 38.0°C rectal or 37.5°C axillary) and one or more of the following signs: neck stiffness, altered consciousness with no other alternative diagnosis, or other meningeal sign such as bulging fontanelle in children under one year of age.
  If a Cerebrospinal fluid (CSF) sample is available and any known aetiologic agent (bacterial or not) has been identified, it is defined as an aetiology confirmed meningitis.
  The incidence rate will be calculated by dividing the number of study participants reporting at least one event over the follow-up period by the total person-time.

SECONDARY OUTCOMES:
Incidence rate of probable meningitis (final classification) | During the entire study period (From Day 0 up to Month 62)
  At the site level, a suspected probable meningitis case based on clinical symptoms and/or signs is defined by the below characteristics:
  CSF sample is available, no bacterial agent has been identified in the CSF, but some abnormalities in the CSF have been detected (such as turbid macroscopic aspect, positive Gram, positive antigen test, pleiocytosis, abnormal glucose or protein levels) or positive blood culture to a bacterial agent.
  The incidence rate will be calculated by dividing the number of study participants reporting at least one event over the follow-up period by the total person-time.
Incidence rates of clinically suspected meningitis (final classification) | During the entire study period (From Day 0 up to Month 62)
  At the site level, a clinically suspected meningitis case based on clinical symptoms and/or signs is defined by the below characteristics:
  * If a CSF sample is available and all examinations are normal at first line laboratory level, or if no CSF sample is available and no alternative diagnosis.
  The incidence rate will be calculated by dividing the number of study participants reporting at least one event over the follow-up period by the total person-time.
Number of meningitis cases identified at site level (first line laboratory) | During the entire study period (From Day 0 up to Month 62)
  At the site level, a suspected meningitis case based on clinical symptoms and/or signs is defined as:
  * A child with sudden onset of fever (> 38.0°C rectal or 37.5°C axillary) and one or more of the following signs: neck stiffness, altered consciousness with no other alternative diagnosis, or other meningeal sign such as bulging fontanelle in children under one year of age.
Incidence rates of cerebral malaria (diagnosed by Rapid Diagnostic Test [RDT] and/or microscopy) | During the entire study period (From Day 0 up to Month 62)
  Cerebral malaria is defined as:
  * Severe Plasmodium falciparum malaria with impaired consciousness (Glasgow coma score < 11 in children ≥ 2 years of age or Blantyre coma score < 3 in children < 2 years of age); And,
  * If malaria with seizure: coma persisting for > 30 min after the seizure.
  * Other treatable causes of coma should be excluded before diagnosing cerebral malaria (e.g. hypoglycaemia, bacterial meningitis).
  Suspected malaria cases routinely tested using RDT will have a blood smear for reading by microscopy in parallel, in order to measure sensitivity and specificity. This is done for all suspected cases presenting at primary health care facilities one day per month during the first year of the study.
  The incidence rate will be calculated by dividing the number of study participants reporting at least one event over the follow-up period by the total person-time.
Incidence rates of malaria episodes diagnosed by RDT and/or microscopy | During the entire study period (From Day 0 up to Month 62)
  Any malaria is uncomplicated malaria (i.e. Plasmodium parasitaemia >0 detected by microscopy and/or RDT, presence of fever (≥37.5°C) reported by parent(s)/LARs or recorded at time of presentation and without severity signs or vital organ dysfunction) and severe malaria (SM) (i.e. P. falciparum parasitaemia >0 detected by microscopy and/or RDT, one/more of the following: impaired consciousness, prostration, multiple convulsions, acidosis, hypoglycemia, severe malarial anemia, renal impairment, jaundice, pulmonary oedema, significant bleeding, shock, hyperparasitemia). Severe vivax malaria is SM but with no parasite density thresholds. Cerebral malaria is SM with impaired consciousness with the exclusion of other treatable causes of coma. The incidence rate will be calculated by dividing the number of subjects reporting at least one event over the follow-up period by the total person-time.
Incidence rates of anaemia cases at hospital entry among hospitalised children | During the entire study period (From Day 0 up to Month 62)
  This outcome measure is assessed for children included only in active surveillance.
  Anaemia is defined as:
  * All anaemia: haemoglobin <11 (grams per decilitre) g/dL.
  * Severe anaemia: haemoglobin <7g/dL. The incidence rate will be calculated by dividing the number of study participants reporting at least one event over the follow-up period by the total person-time.
Incidence rates of hospitalisation cases | During the entire study period (From Day 0 up to month 62)
  Hospitalisation is defined as:
  All causes and hospitalisations for any malaria (including P. falciparum malaria), severe malaria (including P. falciparum malaria) and cerebral malaria.
  A hospitalised study participant with malaria (including P. falciparum malaria) and for whom malaria is the primary cause of hospitalisation.
  This outcome measure is assessed for children included only in active surveillance.
  The incidence rate will be calculated by dividing the number of study participants reporting at least one event over the follow-up period by the total person-time.
Number of deaths | During the entire study period (From Day 0 up to month 62)
  Death is defined as:
  * Malaria attributed death (including P. falciparum malaria) defined as a fatality for which malaria (including P. falciparum malaria) is listed as a contributing cause of death, based on either verbal autopsy using the INDEPTH Standard Verbal Autopsy Questionnaire for children, who died at home or medical judgment/medical records for children who died at a primary health care facility or hospital.
  * Deaths attributed to an AE defined as a fatality for which an AE is listed as a contributing cause of death, based on either verbal autopsy using the INDEPTH Standard Verbal Autopsy Questionnaire for children, who died at home or medical judgment/medical records for children who died at a primary health care facility or hospital.
  The incidence rate (mortality rate) will be calculated by dividing the number of study participants reporting at least one event over the follow-up period by the total person-time.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (5):
- Ghana (2):
  - GSK Investigational Site, Kintampo
  - GSK Investigational Site, Navrongo
- GSK Investigational Site, Kisumu, Kenya
- Malawi (2):
  - GSK Investigational Site, Chikwawa
  - GSK Investigational Site, Mangochi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ndeketa L, Haine V, Debois M, Asante KP, Agyapong PD, Kaali S, Devadiga R, Harrison SBE, Boahen O, French N, Kayan K, Ogutu B, Adeniji E, Kariuki S, Owusu-Agyei S, Olewe F, Jere TM, Maleta K, Mategula D, Mzanga P, Phiri VK, Ansah PO, Orimbo J, Ansah NA, Orsini M, Ong'echa JM, Oduro AR, Sifuna PM, Azongo DK, Otieno W, Bangre O, Kaburise MB, Ababio LO, Oyieko JN, Sing'oei V, Amoit SK, Nyangulu W, Schuerman L, Awuni D, Ochieng BO, Onyango I, Odera-Ojwang P, Oguk EA, Mendoza YG, Cherop RY, Okoth GO, Cravcenco C, Chipatala R, Roman F, Oneko M, Savic M; RTS,S Epidemiology EPI-MAL-003 Study Group. Effectiveness of the RTS,S/AS01E malaria vaccine in a real-world setting over 1 year of follow-up after the three-dose primary schedule: an interim analysis of a phase 4 study in Ghana, Kenya, and Malawi. Lancet Glob Health. 2026 Jan;14(1):e61-e69. doi: 10.1016/S2214-109X(25)00415-2. Epub 2025 Nov 6. PMID 41207319
- [Derived] Haine V, Oneko M, Debois M, Ndeketa L, Agyapong PD, Boahen O, Harrison SBE, Adeniji E, Kaali S, Kayan K, Owusu-Agyei S, French N, Kariuki S, Devadiga R, Ogutu B, Ansah NA, Orsini M, Ansah PO, Maleta K, Ong'echa JM, Phiri VK, Mzanga P, Jere TM, Azongo DK, Mategula D, Orimbo J, Oduro AR, Otieno W, Kaburise MB, Ababio LO, Sifuna PM, Amoit SK, Olewe F, Oyieko JN, Achieng Oguk E, Guerra Mendoza Y, Awuni D, Sing'oei V, Onyango I, Schuerman L, Ochieng BO, Okoth GO, Nyangulu W, Cherop RY, Odera-Ojwang P, Cravcenco C, Chipatala R, Roman F, Savic M, Asante KP. Safety of RTS,S/AS01E malaria vaccine up to 1 year after the third dose in Ghana, Kenya, and Malawi (EPI-MAL-003): a phase 4 cohort event monitoring study. Lancet Glob Health. 2025 Jun;13(6):e995-e1005. doi: 10.1016/S2214-109X(25)00096-8. Epub 2025 Apr 24. PMID 40288377